CLINICAL TRIAL: NCT00908674
Title: Measure of Androcur Effects on Quality of Life at Prostate Cancer Patients
Brief Title: Androcur Effects on Quality of Life
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Hungária Kft.
Other Study IDs: 14166; AC0710HU
Record Dates: First submitted 2009-03-24; First posted 2009-05-27 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyproterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Cyproterone acetate (Androcur)

INTERVENTIONS:
Drug: Cyproterone acetate (Androcur) — The study drug will be administered either as monotherapy or in combination with other interventions (surgical castration or LHRH analogue treatment).
  Daily dosage as monotherapy: 200-300 mg cyproterone acetate. Daily dosage following surgical castration: 100-200 mg cyproterone acetate. Daily dosage in combination with an LHRH-analogue: 100-200 mg cyproterone acetate.
  Administration period: 12 months.

SUMMARY:
Androcur is an antiandrogenic drug, which blocks the action of male sex hormones. Androcur is used for treatment of advanced prostate cancer. This study investigates the effect of Androcur on quality of life of prostate cancer patients who are taking the drug for 12 months

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Inoperable prostate tumor or progradiated after surgery/ irradiation therapy
* Locally advanced tumor or distant metastases is present

Exclusion Criteria:

* Patient not fulfil the recruitment criteria
* Liver disease; Dubin-Johnson syndrome; Rotor syndrome; previous or existing liver tumours (in carcinoma of the prostate only if these are not due to metastases); wasting diseases (with the exception of carcinoma of the prostate); depression; previous or existing thromboembolic processes; diabetes with vascular changes; sickle-cell anaemia.
* As regards patients with prostatic carcinoma who have a history of thromboembolic processes and/or an existing sickle-cell anaemia, or diabetes with vascular changes, the risk:benefit ratio must be considered carefully in each individual case before the use of Androcur

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Quality of life change measured by SF-35 questionnaire | Baseline, after 3, 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Hungary